CLINICAL TRIAL: NCT01579825
Title: Evaluation of the Effect of Buffer on the Immune Response to Oral Poliovirus Vaccine in Bangladesh: a Randomized Controlled Trial
Brief Title: Evaluation of Buffer on Immune Response to Oral Polio Vaccine (OPV) in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00003717
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis | interventions — Buffers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffer (Experimental)
  Interventions: Other: Buffer
- Control (No Intervention)

INTERVENTIONS:
Other: Buffer — 5 ml of oral buffer solution containing 64 mg of sodium bicarbonate plus 24 mg of sodium citrate. The buffer will be administered prior to each dose of OPV at 6, 10 and 14 weeks of age.
  Arms: Buffer

SUMMARY:
Hypothesis:

The immunogenicity of oral polio vaccine (OPV) will be enhanced in Bangladeshi infants who receive bicarbonate buffer at the time of polio immunization.

DETAILED DESCRIPTION:
The investigators will conduct a study to evaluate the impact of administering bicarbonate buffer on the serologic responses to oral polio vaccine (OPV) in Bangladeshi infants.

ELIGIBILITY:
Inclusion Criteria:

* infants who are 4-8 weeks old
* residents of study area

Exclusion Criteria:

* received a blood transfusion or any other blood product (such as immune globulin)
* likely to move out of study area within the next four months
* currently enrolled or planning to enroll in another study
* major congenital malformations
* neurologic disorders
* immunodeficiency

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serologic response | 4 weeks after last dose of OPV
  Serologic response rate for each polio virus serotype (1, 2, and 3) in OPV.

CONTACTS AND LOCATIONS:
Overall Officials: Neal A Halsey, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Sylhet, Bangladesh

REFERENCES:
- [Derived] Chandir S, Ahamed KU, Baqui AH, Sutter RW, Okayasu H, Pallansch MA, Oberste MS, Moulton LH, Halsey NA. Effect of buffer on the immune response to trivalent oral poliovirus vaccine in Bangladesh: a community based randomized controlled trial. J Infect Dis. 2014 Nov 1;210 Suppl 1:S390-7. doi: 10.1093/infdis/jiu378. PMID 25316860